CLINICAL TRIAL: NCT05946122
Title: Effect of Atorvastatin as a Renal Protection in Patients With Systemic Inflammatory Response Syndrome Using Renal Arterial Resistive Index
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, lecturer of anesthesia and pain medicine, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 343/ 8-2022
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Renal Protection
MeSH Terms: interventions — Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Drug: placebo drug
- Active ( Ator) group (Active Comparator)
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — oral atorvastatin for renal protection
  Arms: Active ( Ator) group
Drug: placebo drug — tablet resembles atorvastatin
  Arms: control group

SUMMARY:
Offering renal protection in systemic inflammatory response syndrome by atorvastatin

ELIGIBILITY:
Inclusion Criteria:

* Patients ( male and female) with systemic inflammatory response ( total leucocytic count >12,000 mm3'. temperature >38 C, Heart rate >90 b/min and respiratory rate>20 cycle).

Exclusion Criteria:

* Hemodynamic instability
* Pre-admission chronic kidney disease.
* Intra-vascular coagulopathy
* Patients with myopathy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | one week
  incidence or acute kidney injury

SECONDARY OUTCOMES:
renal resistive vascular index | one week
  renal resistive index
APACHE score ( acute physiology and chronic health evaluation) | one week
  acute physiology and chronic health evaluation, values below 40 are considered normal while values between 41 and 71 are considered abnormal .
length of ICU stay | two weeks
  days of ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Maher Raouf, Minya, Minia University, Egypt